CLINICAL TRIAL: NCT07307300
Title: Risk Stratification of Patients With Non-Visible Hematuria - A Prospective Validation Study Using a Urine Marker-Based Assessment (Xpert® Bladder Cancer Detect)
Brief Title: Study on Risk Assessment for Patients With Microscopic Hematuria (Non-Visible Blood in Urine) Using a Urine Marker Test
Acronym: UroDetect III
Status: Not yet recruiting | Type: Observational
Sponsor: Christian Bolenz (Other)
Collaborators: Cepheid (Industry); Prof. Dr. med. Bernd Schmitz-Dräger (Unknown)
Responsible Party: Sponsor-Investigator, Christian Bolenz, Prof. Dr. med. Christian Bolenz, University Hospital Ulm
Organization: University Hospital Ulm (Other)
Other Study IDs: UroDetect III
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Hematuria
Keywords: Non-visible hematuria; Microscopic hematuria; Bladder cancer risk; Xpert Bladder Cancer Detect; Risk stratification; Diagnostic assessment; Urinary marker
MeSH Terms: conditions — Hematuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this clinical study is to learn how well a urine test called Xpert® Bladder Cancer Detect (Xpert BC-D) can help doctors assess the risk of bladder cancer in people with non-visible blood in their urine (microscopic hematuria). The main questions it aims to answer are:

* Can the Xpert BC-D test accurately identify people at higher risk for bladder cancer?
* Can combining the test results with other clinical information improve risk assessment compared to standard evaluation methods?

Participants will:

* Have leftover urine from the routine initial evaluation tested with the Xpert® Bladder Cancer Detect assay
* Complete questionnaires about urinary symptoms using the modified IPSS and ICIQ-FLUT-S forms
* Attend a first visit for medical evaluation and cystoscopy
* Attend a follow-up visit 3 to 6 months later for additional testing and questionnaires

This study includes adults over 40 years of age who have had microscopic hematuria detected within the past six months. People with a history of bladder cancer, urinary tract surgery, or certain other medical conditions, as well as individuals who are currently pregnant, cannot participate.

The study will be conducted at 20-24 sites in Germany and Austria and will last approximately 27 months, with each participant involved for about 6 months. The results of this study may help doctors better decide which patients need further invasive testing, potentially reducing unnecessary procedures.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form after being informed about the study
* Willing and able to follow the study requirements
* Non-visible blood in the urine, found within the past 6 months
* Age over 40 years

Exclusion Criteria:

* Previous diagnosis of bladder cancer
* Too much protein in the urine (shown by urine test)
* Current urinary tract infection (symptoms like pain or frequent urination, plus bacteria found in urine test)
* Current pain in the urinary tract or lower belly, pain score greater than 2 on a 0-10 scale
* Signs of kidney-related blood in the urine (found by special urine test)
* Bladder examination with a camera (cystoscopy) within the past 12 months
* Pregnancy
* Visible blood in the urine within the past year
* Previous surgery on the urinary tract
* Previous radiation treatment to the pelvic area
* Permanent tube or foreign body in the urinary tract (such as a catheter)
* Participation in another clinical study at the same time or within 30 days before this study
* Detained under legal or official authority
* Medical, psychological, or social problems that would make it hard to follow the study requirements
* Not able to understand the study information well enough to give consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over 40 years with non-visible blood in the urine. Participants are either initially identified by referring primary care physicians and further evaluated at the study sites for possible inclusion, or they are directly identified at the study sites during routine evaluation when microhematuria is detected. Recruitment takes place at multiple urology clinics in Germany and Austria.
Sampling Method: Non-Probability Sample
Enrollment: 1475 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Validating results of a recent metanalysis (UroDetect II) achieving an overall sensitivity of the Xpert BC-D for UCas of >0.70 and a specificity of >0.65 | From enrollment until completion of follow-up at 6 months

SECONDARY OUTCOMES:
Effective detection of high impact tumors (HITs, defined as Ta G3/HG, CIS, and ≥T1 urothelial cancer) | From enrollment until completion of follow-up at 6 months
Validating results from a recent meta-analysis demonstrating improved risk stratification by combining the Xpert BC-D results with clinical parameters | From enrollment until completion of follow-up at 6 months
Simulating application of current major guideline recommendations, a significantly better discrimination between patients at low/high risk for subsequent UCa diagnosis for: The Xpert BC-D results and combinations from Xpert BC-D results and clinical | From enrollment until completion of follow-up at 6 months
Cost-benefit considerations (based on structured information e.g. from GOÄ and EBM) | From enrollment until completion of follow-up at 6 months
Investigating the rate of negative TUR-Bs triggered by standard-of-care (SOC) vs. positive findings by Xpert BC-D results and respective combination with clinical results. (study not powered for confirmation of a significant difference) | From enrollment until completion of follow-up at 6 months
Prospective assessment of symptoms of nvH patients (assessment using modified versions of ICIQ-FLUTS and IPSS) | From enrollment until completion of follow-up at 6 months
Investigating the frequency of conditions requiring medical and/or surgical intervention resulting from nvH assessment | From enrollment until completion of follow-up at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Pediatric Urology University Hospital Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data may be shared upon reasonable request with qualified researchers after publication of the main study results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available from 6 months after publication of the main study results for a period of 5 years.
Access Criteria: Access to individual participant data (IPD) and supporting information will be granted upon reasonable request. Qualified researchers with a methodologically sound proposal and a clear scientific rationale will be eligible to apply for access.
  Approval for data access will be granted by the Sponsor-Investigator in coordination with the Data Protection Officer of the affiliated organization (UHUlm) and, if applicable, in consultation with the responsible Ethics Committee. Requests will be evaluated according to predefined criteria for scientific merit, data protection, and regulatory compliance (e.g., GDPR).
  Approved applicants will be required to sign a Data Use Agreement (DUA) specifying conditions of use, including restrictions on re-identification, redistribution, and secondary use outside the agreed scope. All shared data will be de-identified and will be provided via a secure, controlled-access repository or through secure file transfer, depending on feasibility.